CLINICAL TRIAL: NCT00685620
Title: Reinforcement-Based Treatment and Abstinence-Contingent Housing for Drug Abusers
Acronym: CASA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Maxine Stitzer, Ph.D., Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPR010213-01
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2008-05

CONDITIONS: Drug Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (No Intervention): Standard care following detoxification
- Group 2 (Active Comparator): Recovery housing following detoxification
  Interventions: Behavioral: Reinforcement Based Treatment
- Group 3 (Experimental): Recovery housing plus counseling
  Interventions: Behavioral: Reinforcement Based Treatment

INTERVENTIONS:
Behavioral: Reinforcement Based Treatment — 3 group random assignment to receive standard care, recovery housing alone, or recovery housing plus behavioral treatment
  Arms: Group 2; Group 3

SUMMARY:
Purpose of the project is to examine the effectiveness of Reinforcement-Based Treatment (RBT) on drug abuse and psychosocial outcomes of iner city opiate abusers who have recently completed a brief detoxification.

DETAILED DESCRIPTION:
Participants are randomized into one of 3-groups: 1) those receiving intensive behavioral therapy plus abstinence-contingent housing, 2) those receiving recovery housing alone, and 3) those receiving standard care (referrals to community providers). For the two groups receiving recovery housing, rent payment is provided for a period of 3 months, as long as the participant remains drug-free.

ELIGIBILITY:
Inclusion Criteria:

* opiate dependent agree to live in recovery housing

Exclusion Criteria:

* acute psychiatric disorder pregnant over 65

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2002-08; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Drug abstinence at follow-up | 1, 3 and 6 months

SECONDARY OUTCOMES:
Rates of employment | 1, 3, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Maxine Stitzer, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Tuten M, DeFulio A, Jones HE, Stitzer M. Abstinence-contingent recovery housing and reinforcement-based treatment following opioid detoxification. Addiction. 2012 May;107(5):973-82. doi: 10.1111/j.1360-0443.2011.03750.x. Epub 2012 Feb 28. PMID 22151478